CLINICAL TRIAL: NCT00408122
Title: Evaluation of Positron Emission Tomography/ CT Scan, Endoscopic Ultrasono¬Graphy, and Laparoscopic Ultrasonography in the Preoperative Assess¬Ment of Resectability in Patients With Primary and Secondary Liver Cancer
Brief Title: Evaluation of Preoperative Investigations in Patients With Liver Cancer
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Alan Patrick Ainsworth, dr, Odense University Hospital
Other Study IDs: VF-20060109
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Primary Liver Cancer; Liver Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: PET/CT scan and EUS

SUMMARY:
The aim of the study is to evaluate the diagnostic procedures emission tomography in combination with a CT scan (PET/CT) and endoscopic ultrasonography (EUS) in the preoperative evaluation of resectability of patients with primary or secondary liver cancers.

ELIGIBILITY:
Inclusion Criteria:

* all patients who are referred to The Department of Surgery, Odense University Hospital, for surgical treatment of suspected or biopsy proven primary or secondary liver cancer.

Exclusion Criteria:

* age less than 18 years
* patients who are not fit for liver surgery because of co-morbidity
* patients for whom the extra investigations in the study are considered to give an increased risk because of co-morbidity such as

  * Patients with s-creatinin > 150 micromol/l
  * Patients who take peroral antidiabetic drugs or have a poorly regulated diabetes mellitus
* patients who do not understand the patient information
* patients who do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAtients with liver tumors
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning O Nielsen, MD, DMsc, Principal Investigator — dept. of Surgery, Odense University Hospital
Locations (1):
- Dept of Surgery, Odense university Hospital, Odense, Denmark